CLINICAL TRIAL: NCT00480506
Title: Monitoring of Erythroid Lineage Specific Chimerism Following Allogeneic Hematopoietic Transplantation for Thalassemia Major
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Catherine Wu, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 04-078
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Thalassemia Major
Keywords: chimerism; allogenic hematopoietic transplantation; assay
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect peripheral blood and bone marrow aspirate samples from thalassemia patients in Tehran, in a collaborative effort to develop an erythroid lineage specific chimerism assay applicable to patients with thalassemia. Development of such an assay would be useful both for identification of the exact mutation causing the disease, as well as for providing a direct method to measure and monitor the kinetics of donor erythropoiesis in this patient population following transplant.

DETAILED DESCRIPTION:
* In the first phase of the study we will develop a panel of reagents designed to identify predominant thalassemia mutations in the Iranian population, as well as alternative highly variable erythroid specific polymorphisms. To determine how informative this panel is, these reagents will be applied to samples collected from patients homozygous for the disorder, and compared to patients with thalassemia trait and normal Iranian donors.
* In the second phase, we propose to serially measure and compare erythroid lineage chimerism with overall genomic chimerism following transplant. Samples will be collected from participants before and at 1, 2, 3, 6 and 12 months following transplant and cryopreserved. Peripheral blood from the stem cell donor will also be collected and cryopreserved. Participants will undergo myeloablative or nonmyeloablative transplant.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia patients being treated at Shariati Hospital in Tehran.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thalassemia patients being treated at Shariati Hospital in Tehran.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2004-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Wu, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States
- Tehran University of Medical Sciences, Tehran, Iran